CLINICAL TRIAL: NCT01627353
Title: Post Hysterectomy Pain Prevention: Randomized Clinical Trial of High Volume Preoperative Wound Infiltration and Pain Specific Anesthetic Protocol Versus Standard of Care (no Wound Infiltration and Routine Anesthetic Protocol)
Brief Title: Post Hysterectomy Pain Prevention: Pre-op Wound Infiltration With Anesthetic Protocol Versus Standard of Care
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Wynne Innez Leung, Clinical Assistant Professor, General, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-23700
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Hysterectomy
Keywords: Hysterectomy; Pain Prevention; Wound Infiltration
MeSH Terms: interventions — Standard of Care; Magnesium Sulfate; Dexamethasone; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Current Standard of Care at Rockyview General Hospital for Post Hysterectomy Pain Prevention(no wound infiltration and routine anesthetic protocol).
  Interventions: Procedure: Standard of care
- Pre-emptive wound infiltration (Experimental): The Wound Infiltration Group will receive 100 mL 0.25% marcaine plain distributed as follows: 50 mL subcutaneously prior to skin incision along entire length of planned incision line, 50 mL subfascially prior to fascial incision, with 10 mL infiltrated directly into the rectus muscles bilaterally.
  Interventions: Procedure: Pre-emptive wound infiltration

INTERVENTIONS:
Procedure: Standard of care — Current Standard of Care at Rockyview General Hospital for Post Hysterectomy Pain Prevention(no wound infiltration and routine anesthetic protocol).
  Arms: Standard of Care
Procedure: Pre-emptive wound infiltration — The Wound Infiltration Group will receive 100 mL 0.125% marcaine plain distributed as follows: 50 mL subcutaneously prior to skin incision along entire length of planned incision line, 50 mL subfascially prior to fascial incision, with 10 mL infiltrated directly into the rectus muscles bilaterally.
  The Anesthetic will be given as determined appropriate to the patient by the staff anesthetist with the addition of the following: 2 grams of Magnesium Sulphate, 10 mg of Dexamethasone, and 3 mg/kg of Lidocaine, half of which is given on induction and half of which is infused throughout the remainder of the case.
  Other Names: Magnesium Sulphate; Dexamethasone; Lidocaine
  Arms: Pre-emptive wound infiltration

SUMMARY:
The study is a blinded randomized clinical trial, comparing policies of high volume preemptive wound infiltration with a specific anesthetic cocktail versus standard of care (no wound infiltration and routine anesthesia) for post operative pain management after hysterectomy. Morphine use and pain will be measured during index admission, and pain will also be measured six weeks postoperatively. The study will be conducted at a single site, Rockyview General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* women may be included if they require total abdominal hysterectomies (+/- BSO) at Rockyview hospital.

Exclusion Criteria:

* have endometrial cancer,
* require a vertical midline incision,
* have any additional surgery planned
* have a contraindication to morphine, Magnesium Sulfate, Dexmethasone, Lidocaine or Marcaine
* have difficulty communicating in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Post Operative Morphine | For the entire post-operative hospital admission (3 days on average)
  The amount of post operative morphine (PCA IV) will be recorded from the PCA device each day by the Acute Pain Service Nurses. The total dose (mg morphine) will be recorded for each 24 hour period, and summed for the complete postoperative period of admission.

SECONDARY OUTCOMES:
Pain measurement using Visual Analogue Scale (VAS) post operatively | Daily until discharge (3 days on average)
  Patients will complete pain VAS in recovery and each hospital day post operatively until discharge.
  The majority of papers comparing acute postoperative pain use a VAS. It is a simple measure that is easy to use by patients and currently in use by nurses at our site both in the post anesthetic recovery room and on the units. The VAS measures patient perceived pain intensity on a 10cm single axis scale ranging from no pain (0 cm) to worst pain ever experienced (10cm).
Time in recovery (hours) | Until discharge from recovery (on average 2 hours)
  Time in recovery (hours): will be collected from the recovery room chart.
Morphine use in recovery | Until discharge from recovery (on average 2 hours)
  Morphine use in recovery (mg of morphine): will be collected from the recovery room chart.
Adverse events as a result of morphine overdosage | Until discharge from recovery (on average 2 hours)
  Any emergencies as a result of morphine overdosage: will be collected from the recovery room chart.
Change in pain score | baseline - 6 weeks post-operative
  Change in pain score: will be calculated as: baseline SF-MPQ2 minus six week SF-MPQ2 for total and each subscore of SF-MPQ2.

CONTACTS AND LOCATIONS:
Overall Officials: Wynne Leung, Principal Investigator — University of Calgary
Locations (1):
- Rockyview General Hospital, Calgary, Alberta, Canada